CLINICAL TRIAL: NCT05122910
Title: Assessing the Implementation and Feasibility of the Stress Management and Resilience Training - Moral Resilience Program (SMART-MR) With Frontline Clinical Staff at The Ottawa Hospital: A Non-randomized Pilot Study
Brief Title: Assessing the Implementation and Feasibility of the SMART-MR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Edward Spilg, Assistant Professor, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20210559-01H
Record Dates: First submitted 2021-10-22; First posted 2021-11-17 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Moral Injury
Keywords: Moral Distress; Moral Resilience; Healthcare workers; COVID-19
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART-MR Program (Experimental): Participants will participate in the Stress Management and Resilience Training - Moral Resilience (SMART-MR) program.
  Interventions: Behavioral: Stress Management and Resilience Training - Moral Resilience (SMART-MR) program

INTERVENTIONS:
Behavioral: Stress Management and Resilience Training - Moral Resilience (SMART-MR) program — All participants will attend an initial 2.5 hour workshop and a 1-hour follow-up workshop. The workshop will include general resilience strategies with a focus on the moral/ethical dimensions of clinical practice to offer participants specific skills to address ethical challenges. In addition to the workshops, there will be follow-up supplemental resources.

SUMMARY:
The objective of the proposed pilot study is to assess the feasibility and implementation of the SMART-MR program, an integration of stress management, general resilience, and moral resilience skills, with frontline staff who provide direct patient care at The Ottawa Hospital (TOH).

DETAILED DESCRIPTION:
Many of the sources of stress facing healthcare workers during the COVID-19 pandemic involve difficult ethical trade-offs that give rise to moral distress. Moral distress has personal consequences for healthcare workers, notably for their mental health, and wider consequences for the organization and health system as a whole as it negatively affects quality of care, patient satisfaction, and the recruitment, retention and satisfaction of staff. Moral resilience refers to the capacity of an individual to sustain or restore their integrity in response to moral adversity and has been raised as a potential way to mitigate moral distress.

The Stress Management and Resilience Training (SMART) program is one of the few evidence-based interventions designed to build resilience in healthcare workers. The SMART program is a brief, neuroscience-based intervention, typically delivered in a single 90-minute session. The structured program teaches self-care skills by developing intentional attention and the ability to reframe potentially stressful situations more quickly.

Recently, a modified version of the existing SMART program, SMART-Moral Resilience (SMART-MR), has been developed with an additional focus on reducing moral distress and building moral resilience for healthcare workers. The synergy of general resilience strategies with focus on the moral/ethical dimensions of clinical practice offer clinicians specific skills to address ethical challenges. We believe implementing the SMART-MR program with frontline staff during the COVID-19 pandemic is warranted. Therefore, we plan to pilot this innovative intervention at TOH to assess its feasibility and implementation.

ELIGIBILITY:
Inclusion Criteria:

• full-time or part-time TOH staff who provide direct patient care, including: attending physicians, nurses, allied health, social workers and spiritual care providers

Exclusion Criteria:

• TOH staff members who do not provide direct patient care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Change in the Measure of Moral Distress-Health Professionals (MMD-HP) | Baseline, 12 weeks follow-up
  27-item scale that measures healthcare professionals' current levels of moral distress. Respondents rate each item on two Likert scales to indicate: how often a situation occurs during their practice (frequency: 0 = never, 4= very frequent) and how distressing it is when it occurs (distressing: 0= none, 4= very distressing). The frequency score (f) is multiplied by the distress score (d) to receive a composite score ("fxd", range 0-16). These scores are summed to create the overall MMD-HP score (ranging from 0-432), with higher scores indicative of higher moral distress.
Change in the Rushton Moral Resilience Scale (RMRS) | Baseline, 12 weeks follow-up
  17-item scale assessing moral resilience in healthcare workers. Respondents rate their level of agreement with each item on a Likert scale from 1 ("disagree") to 4 ("agree"). The items form 4 factors: 1) response to moral adversity; 2) personal integrity; 3) relational integrity; and 4) moral efficacy and a total summative score is calculated.

SECONDARY OUTCOMES:
Change in the Maslach Burnout Inventory-2 item version (MBI-2 item) | Baseline, 12 weeks follow-up
  2 items that capture the emotional exhaustion (i.e., "I feel burned out from my work") and depersonalization (i.e., "I have become more callous toward people since I started this job") domains of burnout. Respondents rate their level of agreement with these items on a scale from 0 (never) to 6 (everyday). A score of >3 on either item is considered indicative of burnout.
Change in the Perceived Stress Scale-10 item (PSS-10) | Baseline, 12 weeks follow-up
  10-item scale that provides a global measure of perceived stress. Responses range on a 5-point scale from "never" to "very often." A higher score indicates greater stress.
Change in the Generalized Anxiety Disorder 7-item (GAD-7) scale | Baseline, 12 weeks follow-up
  7-item questionnaire that assessed generalized anxiety. Response options are "not at all," "several days," "more than half the days," and "nearly every day," scored as 0, 1, 2, and 3, respectively. Cut-off scores of 5, 10, and 15 delineate mild, moderate, and severe anxiety, respectively; scores ≤4 correspond to minimal anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Spilg, MBChB, Principal Investigator — University of Ottawa
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No